CLINICAL TRIAL: NCT06382558
Title: Evaluating Validity and Reliability of a Novel In-house Developed, Robot-based Sensorimotor Processing Assessment Paradigm for the Upper Limb in the Chronic Phase After Stroke.
Brief Title: Validity and Reliability of Sensorimotor Processing Paradigm
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Prof Geert Verheyden, Prof. Dr. Geert Verheyden, KU Leuven
Other Study IDs: s68470; C2M/23/060 (Other Grant/Funding Number: KU Leuven)
Record Dates: First submitted 2024-04-18; First posted 2024-04-24 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Stroke
Keywords: Stroke; Upper limb; Somatosensation; Sensory processing; Robotic assessment; Kinematics
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Chronic stroke patients: Patients who experienced a first unilateral stroke at least 6 months ago
- Healthy controls: Healthy subjects with no history of any neurological condition and who are in the same age group as the chronic stroke patients

SUMMARY:
Sensorimotor function of the upper limb is often impaired after stroke, even in the chronic phase (minimum 6 months after stroke). Currently, an optimal assessment for sensory processing, one of the most important sensory functions, does not exists. However, our research team has developed a novel assessment paradigm using the KINARM End-Point robot to assess the level of sensory processing of the upper limb. Within a previous study, the investigators examined the validity within 20 chronic stroke patients and 80 age-matched healthy controls by comparing the novel robotic assessment with a set of existing clinical and robotic assessments for the upper limb. The investigators hypothesize that the stroke patients will show a poorer performance on this novel assessment compared to the healthy controls, that the novel assessment will show better correlation coefficients with other sensory tests compared to motor tests, that the novel assessment can differentiate between different motor subgroups of chronic stroke patients, and that the novel assessment shows good test-retest reliability.

DETAILED DESCRIPTION:
Sensorimotor function of the upper limb is often impaired after stroke, even in the chronic phase (minimum 6 months after stroke). These impairments may lead to significant limitations in activities of daily living and may negatively affect quality of life. It is therefore of importance to accurately assess upper limb impairments. Clinical assessments exist for both motor and somatosensory function, but lack good psychometric properties. Robotics show promising potential and is readily available to assess motor function and proprioception. Robotic assessment for sensory processing is currently not yet available, despite being the most relevant somatosensory function. Indeed, sensory processing shows the strongest association with upper limb movement, and only shows incomplete recovery at 6 months after stroke.

Within a previous study of our research team, a novel robotic assessment of sensory processing was developed, using the Kinarm End-Point Lab (BKIN Technologies Ltd., Canada). That study was set up to initially validate this novel robotic assessment and to collect pilot data to form the basis for future research. 20 chronic stroke patients and 80 age-matched controls underwent extensive clinical and robotic assessment of upper limb motor and somatosensory function. For the cross-sectional study, the investigators aim to build further on this previous research. By recruiting 60 additional chronic stroke patients and combining both data of the previous study and this study, the investigators aim to examine the validity and reliability of this novel assessment in a bigger and more heterogeneous group of chronic stroke participants. The investigators hypothesize that stoke patients have a worse performance on this novel robotic assessment compared to healthy controls, that the novel assessment correlates more to standard sensory assessments compared to standard motor assessments, that the novel assessment can differentiate between motor subgroups of chronic stroke patients, and that the novel assessment shows good test-retest reliability.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained prior to any screening procedures
2. First-ever unilateral, supra-tentorial stroke (as defined by WHO)
3. At least 18 years old
4. Being in the chronic phase after stroke (i.e. being at least 6 months after stroke)
5. Motor impairment in the upper limb, defined as Fugl-Meyer score >22 out of 66 to demonstrate moderate to full upper limb motor function (patients scoring <23 out of 66 will not be able to comply with the KINARM protocol)

Exclusion Criteria:

1. Any serious musculoskeletal and/or other neurological disorders
2. Severe communication or cognitive deficits that interfere with the protocol
3. Any disorder, which in the investigator's opinion might jeopardise participant's safety or compliance with the CIP.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All participants will be recruited from the community sample
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2024-04-10 (Actual); Primary Completion 2025-03-19 (Actual); Study Completion 2025-03-19 (Actual)

PRIMARY OUTCOMES:
Kinarm: Passive and active discrimination task | up to 2 days
  Newly-developed task on the Kinarm End-Point Lab used to assess passive and active sensory processing

SECONDARY OUTCOMES:
Kinarm: Arm position matching task | 1 day
  Assessment of limb position sense using a 9-target mirror-matching task on the Kinarm End-Point Lab
Kinarm: Visually guided reaching task | 1 day
  Assessment of motor function using a 4-target centre-out reaching task on the Kinarm End-Point Lab
Erasmus modified Nottingham sensory assessment | 1 day
  Clinical assessment of sensory processing with an area under the curve based scoring system, with higher scores meaning better performance
Tactile discrimination test | 1 day
  Clinical assessment of sensory processing with an area under the curve based scoring system, with higher scores meaning better performance
Tactile functional object recognition | 1 day
  Clinical assessment of sensory processing on an ordinal scale ranging from 0 to 42, with higher scores meaning better performance
Stereognosis section of the original Nottingham sensory assessment | 1 day
  Clinical assessment of sensory processing on an ordinal scale ranging from 0 to 22, with higher scores meaning better performance
Wrist position sense test | 1 day
  Clinical assessment of wrist position sense on a continuous scale, with lower scores meaning better performance
Perceptual threshold of touch | 1 day
  TENS-based assessment of exteroception on a continuous scale, with lower scores meaning better performance
Fugl-Meyer upper extremity assessment | 1 day
  Clinical assessment of motor function on an ordinal scale ranging from 0 to 66, with higher scores meaning better performance
Action research arm test | 1 day
  Clinical assessment of motor activity performance on an ordinal scale ranging from 0 to 57, with higher scores meaning better performance
Barthel index | 1 day
  Clinical assessment of activities of daily living on an ordinal scale ranging from 0 to 20, with higher scores meaning better performance
Montreal cognitive assessment | 1 day
  Clinical assessment of cognitive function on an ordinal scale ranging from 0 to 30, with higher scores meaning better performance
Star cancellation test | 1 day
  Clinical assessment of visuospatial neglect on an ordinal scale ranging from 0 to 54, with higher scores meaning better performance, and a score below 44 indicating the presence of visuospatial neglect

CONTACTS AND LOCATIONS:
Overall Officials: Geert Verheyden, Principal Investigator — KU Leuven
Locations (1):
- KU Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided